CLINICAL TRIAL: NCT03205579
Title: Effectiveness of Pain Education to Improve Cancer Pain Management in Hospitalized Patients
Brief Title: Pain Education to Improve Cancer Pain Management Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si231/2017
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Pain; Inpatient; Cancer
MeSH Terms: conditions — Pain; Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video group (Experimental): Video cancer pain education (10 minutes ) the knowledge includes cancer pain definition, cancer pain treatment, pain assessment and role of patient in cancer pain management.
  Interventions: Other: Video group
- Conventional group (Active Comparator): Face to face cancer pain education by trained nurse (10 minutes)the knowledge includes cancer pain definition, cancer pain treatment, pain assessment and role of patient in cancer pain management.
  Interventions: Other: conventional group

INTERVENTIONS:
Other: Video group — Using video for educate cancer pain patients
  Arms: Video group
Other: conventional group — Face to face cancer pain education by trained nurse
  Arms: Conventional group

SUMMARY:
Cancer pain is one of the problems of treating cancer pain. Although, there is a WHO analgesic ladder to improve this problem, it is still inadequate pain control. Pain does not affect only physical but also emotional and quality of life.

From review literatures we found that patients' knowledge about cancer pain management is inaccurate; for example, fear to use opioid, try to patience of pain, concerning only cancer treatments, which can cause of unfavorable pain management outcome.

Therefore, we will conduct the RCT of using pain education by video comparing to conventional face to face pain education by nurse in hospitalized cancer pain patients.We will use 25 MCQs examination for testing pre-post intervention to test level of understanding of patients. The measurements are NRS, ThaiHADs and FACT-G at the first and last day of study. We expect that NRS should improve more than 50% at the seven day of study.

DETAILED DESCRIPTION:
protocol Randomized controlled trial study Sample size is 70 patients divided to 2 groups (35 for video group and 35 for conventional face to face group) Inclusion criteria

1. patients' age 18-70 years old
2. moderate to severe cancer pain
3. ECOG(Eastern cooperative Oncology Group) performance status <= 3
4. Patients can write and read Thai language Exclusion criteria

1.Clinical unstability 2.Confusion and delirium 3.Bed ridden 4.Psychotic problem We will randomly allocate patients by using computer program nQuery advice 6.0. After patients sign inform consent we will record baseline characteristics, assess baseline Numerical rating scale (NRS), emotional status (ThaiHADs), Quality of life status (FACT-G). All patients will do the 25 MCQs test within 30 minutes before intervention. Video group will watch video 10 minutes and conventional group will receive pain education from trained nurse in the same period. The knowledge includes cancer pain definition, cancer pain management, pain assessment and role of patients in cancer pain management. After finishing intervention patients will the same 25 MCQs test (30 minutes) and patients can ask questions to the trained nurse.

All patients will be educated to record pain diary everyday for seven days. All patients will receive standard pain management from the physicians. At the day seven we will assess NRS, ThaiHADs and FACT-G and finish the study.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe pain (NRS>4) cancer pain
* ECOG (Eastern cooperative Oncology group) performance status <=3
* Can read, listen, write Thai language

Exclusion Criteria:

* Clinical instability
* Confusion and delirium
* Bed ridden
* Psychotic problem

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Pain intensity | seven days
  The pain reduction will be assessed and compared using numerical rating (NRS) from 0-10; 0 designating "no pain" and 10 designating " worst possible pain" scale between the first day and the seventh day of study

SECONDARY OUTCOMES:
Emotional status | seven days
  The emotional status of participants will be assessed and compared using Thai-HADs (Hospital Anxiety and Depression scale) between the first day and the seventh day of study. The score will be analyzed into depression and anxiety. the score 0-7 for either sub scale being in normal range, 8-10; being just suggestive of the presence of the respective state, a score of 11 or higher indicating probable presence of the mood disorder(Depression and Anxiety).
Functional assessment | seven days
  Functional status will be assessed and compared using FACT-G between the first day and the seventh day of study. The subscale including physical well-being, social/family well-being, emotional well-being and functional well-being. Each items scored from 0-4; from 0 means "not at all" to 4 means "very much". The higher score would indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Suratsawadee Wangnamthip, md, Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (2):
- Thailand (2):
  - Faculty of medicine Siriraj Hospital Mahidol University, Bangkoknoi, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wangnamthip S, Euasobhon P, Siriussawakul A, Jirachaipitak S, Laurujisawat J, Vimolwattanasarn K. Effective Pain Management for Inpatients at Siriraj Hospital: A Retrospective Study. J Med Assoc Thai. 2016 May;99(5):565-71. PMID 27501612
- [Result] van den Beuken-van Everdingen MH, de Rijke JM, Kessels AG, Schouten HC, van Kleef M, Patijn J. Prevalence of pain in patients with cancer: a systematic review of the past 40 years. Ann Oncol. 2007 Sep;18(9):1437-49. doi: 10.1093/annonc/mdm056. Epub 2007 Mar 12. PMID 17355955
- [Result] Yates P, Dewar A, Edwards H, Fentiman B, Najman J, Nash R, Richardson V, Fraser J. The prevalence and perception of pain amongst hospital in-patients. J Clin Nurs. 1998 Nov;7(6):521-30. doi: 10.1046/j.1365-2702.1998.00192.x. PMID 10222947
- [Result] Gureje O, Von Korff M, Simon GE, Gater R. Persistent pain and well-being: a World Health Organization Study in Primary Care. JAMA. 1998 Jul 8;280(2):147-51. doi: 10.1001/jama.280.2.147. PMID 9669787